CLINICAL TRIAL: NCT01777685
Title: Therapeutic Drug Monitoring and Pharmacokinetic Compartmental Analysis of Sulpiride
Brief Title: Therapeutic Drug Monitoring and Pharmacokinetic Compartmental Analysis of Sulpiride After Oral Administration to Healthy Volunteers
Acronym: SUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PPT3
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Sulpiride; Therapeutic drug monitoring; Pharmacokinetics
MeSH Terms: interventions — Sulpiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sulpiride 50 mg (Other)
  Interventions: Drug: Sulpiride

INTERVENTIONS:
Drug: Sulpiride
  Other Names: Dogmatil

SUMMARY:
The present study was adopted to evaluate the pharmacokinetics of sulpiride after oral administration.

DETAILED DESCRIPTION:
The present study was adopted to evaluate the pharmacokinetics of sulpiride after administration of single oral doses of 50 mg in an open-label, one-way study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and not more than 45 healthy male volunteers
* Actual weight no more than ± 30% from ideal body weight based on sex, height, and body frame
* Who had passed all the screening parameters
* Free of any drug exposure known to interfere with the pharmacokinetics or assay of sulpiride for at least 10 days prior to the study
* Who had to be able to communicate effectively with study personnel, be literate, and able to give consent.

Exclusion Criteria:

* A clinically significant abnormal physical exam, medical history, or laboratory studies If they showed a sitting SBP of >140 or <100 mmHg, DBP > 90 or <60mm Hg, or a pulse rate of > 95 or < 50 beats/min at screening A history of serious intolerance, allergy, or sensitivity to fexofenadine The use of any prescription drug within the previous month or use of any over-the-counter medication (with the exception of acetaminophen) within the past 14 days A history of blood dyscrasias A history of alcohol or drug abuse within the past year Donation of blood during the 8 weeks prior to the study or plans to donate blood during or within 8 weeks of completing the study Unable to tolerate vein puncture and multiple blood samplings Any surgical/medical condition that might alter drug absorption, distribution, metabolism, or excretion Cannot follow instructions, in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
•Assessment of the bioequivalence of the oral suspension formulation, the oral solution formulation, and the marketed tablet formulation of levofloxacin, on Days 1, 2, and 3, using the marketed tablet as the reference. Pharmacokinetics of sulpiride | The pharmacokinetic analysis is done after blood sampling
  Assessment of the pharmacokinetics using compartmental and non compartmental analysis of sulpiride after oral administration

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutics Department, Faculty of Pharmacy, Damanhour University, Damanhur, Egypt

REFERENCES:
- [Derived] Helmy SA. Therapeutic drug monitoring and pharmacokinetic compartmental analysis of sulpiride double-peak absorption profile after oral administration to human volunteers. Biopharm Drug Dispos. 2013 Jul;34(5):288-301. doi: 10.1002/bdd.1843. Epub 2013 May 19. PMID 23585286